CLINICAL TRIAL: NCT01828333
Title: Treatment of Severe Malaria - An Operational Comparative Study Between Quinine and Artesunate for the Treatment of Severe Malaria in Hospitals and Health Centers of Kinshasa and Lower Congo
Brief Title: Malaria Treatment With Injectable ArteSunate
Acronym: MATIAS
Status: Completed | Type: Observational
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Other Study IDs: Swiss TPH P 001-01-12
Record Dates: First submitted 2013-03-14; First posted 2013-04-10 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Severe Malaria
Keywords: Malaria; Severe; Artesunate; Quinine; Democratic Republic of Congo
MeSH Terms: conditions — Malaria; Lymphoma, Follicular

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intravenous artesunate - new routine in DRC: 350 patients to be enrolled
  A first study group with the currently used standard for treatment of severe malaria in the DRC, i.v. quinine, was enrolled from 21 October 2012 to 15 January 2013. This study was initially planned as limited scope implementation study with pure observational character (routine diagnosis and treatment, time and motion study, feasibility assessment and costing) and thus not registered. Due to additional publications on i.v. artesunate, non-routine testing for hemoglobin levels before and after treatment plus non-routine follow up was added: Registration of study at this point.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The MATIAS study aims to demonstrate through limited scope implementation studies how injectable artesunate may be progressively rolled out nationwide in the Democratic Republic of the Congo as the preferred treatment for severe malaria.

DETAILED DESCRIPTION:
In 2010 the AQUAMAT study demonstrated that the treatment of severe malaria with artesunate in children reduced the case fatality substantially. An overall reduction of 22.5 % of mortality in African children (< 15 years) was reported using injectable artesunate compared to injectable quinine for treatment of severe malaria caused by Plasmodium falciparum. These results with high quality evidence led to a change in the WHO guidelines for the treatment of severe malaria in 2011. The WHO now recommends intravenous artesunate as the treatment of choice for severe malaria in children and adults. In early 2012 the Programme National de Lutte contre of Paludisme (PNLP) of the DRC with support from the relevant ministry departments decided to follow the WHO guidelines and changed the policy for the treatment of severe malaria in children and adults from injectable quinine to injectable artesunate. However, this process is a complex undertaking, requiring many operational and clinical adaptations. In order to support this process, there is a need for on-site operational information on the process and consequences of the switch from quinine to artesunate. The MATIAS study aims to demonstrate through limited scope implementation studies how injectable artesunate may be progressively rolled out nationwide in the Democratic Republic of the Congo as the preferred treatment for severe malaria.

ELIGIBILITY:
Inclusion Criteria:

Patients (= 2 months old) admitted to one of the study sites and treated for severe malaria with IV quinine in the first part of the study and patients treated with IV/IM artesunate in the second part of the study will be included. Patients need to fulfill the WHO criteria for severe malaria and must be unable to take oral treatment (WHO, 2010, WHO, 2011). In addition all participants need to give their informed consent

Conditions: Positive rapid diagnostic test (RDT) for Plasmodium falciparum HRP2 or lactate dehydrogenase and/or a positive blood slide (thick smear). Patient will be considered to be positive if one of the two tests is positive. In case of negative result of both tests, the patient will not be enrolled in the study and will receive care according to the usual routine practice in the hospital/health center in question.

Definition of severe malaria according to WHO (WHO, 2010): In a patient with P. falciparum asexual parasitaemia and no other obvious cause for the symptoms, the presence of one or more of the following clinical or laboratory features classifies the patient as suffering from severe malaria:

Clinical features (hospitals and health centers):

* impaired consciousness or unrousable coma
* prostration, i.e. generalized weakness so that the patient is unable walk or sit up without assistance
* failure to feed
* multiple convulsions - more than two episodes in 24 h
* deep breathing, respiratory distress (acidotic breathing)
* circulatory collapse or shock, systolic blood pressure < 70 mm Hg in adults and < 50 mm Hg in children
* clinical jaundice plus evidence of other vital organ dysfunction

Complementary Laboratory findings (hospitals only)

* severe anaemia (Hb < 5g/dl, packed cell volume < 15%)
* hypoglycemia (blood glucose < 2.2 mmol/l or < 40 mg/dl)
* metabolic acidosis (plasma bicarbonate < 15 mmol/l)
* serum creatinine > 265 ìmol/l suggesting renal impairment

Exclusion Criteria:

Patients with known serious adverse reactions to quinine and artemisinin derivatives or patients who have received adequate antimalarial treatment 24 hours before admission will not be included in the study.

Women with known or suspected pregnancy in all trimesters will not be included in the study and will be treated with quinine infusions according to the new national DRC guidelines (Programme Nationale de Lutte contre le Paludisme, 2012). According to current routine procedures determination of pregnancy will be done by medical anamnesis and/ or by a positive pregnancy test.

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with severe malaria will be enrolled in four hospitals and five health centers located in four health zones of the Democratic Republic of the Congo, three rural and one urban.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Duration of hospitalization (from registration to discharge) | 3-7 days

OTHER OUTCOMES:
Clinical assessment | 28 days
  * Time from start of IV/IM treatment to initiation of oral treatment
  * Parasite clearance time
  * Clinical status at discharge
  * Signs for tiredness and breathlessness at follow up
Laboratory assessment (exploratory - (see explanation in 1.1.4) | 28 days
  - Hemoglobin nadir during follow up period of 28 days
Time and motion study | 28 days
  - Cumulative staff time required for all steps of patient management, including drug administration
Feasibility and acceptability study | 28 days
  * Perceived feasibility of patient management (as assessed and graded by provider questionnaire)
  * Perceived ease of application of drug treatment (as assessed and graded by provider questionnaire)
  * Perceived quality of case management (including perceived adverse effects) by patient / caretaker (as assessed through patient / caretaker questionnaire)
Analysis of financial cost | 28 days
  - Total financial cost of patient management including treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christian Burri, PhD, Principal Investigator — Swiss Tropical & Public Health Institute; Antoinette Tshefu, MD, Principal Investigator — Kinshasa School of Public Health
Locations (9):
- Democratic Republic of the Congo (9):
  - Centre de Santé CECO, Kimpese, Bas-Congo Province
  - Centre de Santé la Famille, Kimpese, Bas-Congo Province
  - Hôpital Général de Référence IME, Kimpese, Bas-Congo Province
  - Centre de Santé Ngeba, Kisantu, Bas-Congo Province
  - Hôpital Saint Luc de Kisantu, Kisantu, Bas-Congo Province
  - Centre Hospitalier Roi Baudoin 1er Masina, Kinshasa, Kinshasa City
  - Centre de Santé Bita, Maluku, Kinshasa City
  - Centre de Santé Menkao, Maluku, Kinshasa City
  - Centre Hospitalier d'État de Maluku, Maluku, Kinshasa City

REFERENCES:
- [Background] Dondorp AM, Fanello CI, Hendriksen IC, Gomes E, Seni A, Chhaganlal KD, Bojang K, Olaosebikan R, Anunobi N, Maitland K, Kivaya E, Agbenyega T, Nguah SB, Evans J, Gesase S, Kahabuka C, Mtove G, Nadjm B, Deen J, Mwanga-Amumpaire J, Nansumba M, Karema C, Umulisa N, Uwimana A, Mokuolu OA, Adedoyin OT, Johnson WB, Tshefu AK, Onyamboko MA, Sakulthaew T, Ngum WP, Silamut K, Stepniewska K, Woodrow CJ, Bethell D, Wills B, Oneko M, Peto TE, von Seidlein L, Day NP, White NJ; AQUAMAT group. Artesunate versus quinine in the treatment of severe falciparum malaria in African children (AQUAMAT): an open-label, randomised trial. Lancet. 2010 Nov 13;376(9753):1647-57. doi: 10.1016/S0140-6736(10)61924-1. Epub 2010 Nov 7. PMID 21062666
- [Background] Dondorp A, Nosten F, Stepniewska K, Day N, White N; South East Asian Quinine Artesunate Malaria Trial (SEAQUAMAT) group. Artesunate versus quinine for treatment of severe falciparum malaria: a randomised trial. Lancet. 2005 Aug 27-Sep 2;366(9487):717-25. doi: 10.1016/S0140-6736(05)67176-0. PMID 16125588
- [Background] Lubell Y, Riewpaiboon A, Dondorp AM, von Seidlein L, Mokuolu OA, Nansumba M, Gesase S, Kent A, Mtove G, Olaosebikan R, Ngum WP, Fanello CI, Hendriksen I, Day NP, White NJ, Yeung S. Cost-effectiveness of parenteral artesunate for treating children with severe malaria in sub-Saharan Africa. Bull World Health Organ. 2011 Jul 1;89(7):504-12. doi: 10.2471/BLT.11.085878. Epub 2011 Apr 28. PMID 21734764
- [Background] Centers for Disease Control and Prevention (CDC). Published reports of delayed hemolytic anemia after treatment with artesunate for severe malaria--worldwide, 2010-2012. MMWR Morb Mortal Wkly Rep. 2013 Jan 11;62(1):5-8. PMID 23302816
- [Derived] Ferrari G, Ntuku HM, Burri C, Tshefu AK, Duparc S, Hugo P, Mitembo DK, Ross A, Ngwala PL, Luwawu JN, Musafiri PN, Ngoie SE, Lengeler C. An operational comparative study of quinine and artesunate for the treatment of severe malaria in hospitals and health centres in the Democratic Republic of Congo: the MATIAS study. Malar J. 2015 May 30;14:226. doi: 10.1186/s12936-015-0732-1. PMID 26024661